CLINICAL TRIAL: NCT03293576
Title: Integrating Health Psychology Into Hepatitis c Treatment: a Self-efficAcy Intervention to reDuce Injecting Risk behAviour and hePatitis c reinfecTion Rates
Brief Title: A Self-efficAcy Intervention to reDuce Injecting Risk behAviour and hePatitis c reinfecTion Rates
Acronym: ADAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: NHS Tayside (Other Government)
Responsible Party: Principal Investigator, John Dillon, Professor, University of Dundee
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2017PZ04
Record Dates: First submitted 2017-09-05; First posted 2017-09-26 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Hepatitis C
Keywords: Behavioural Medicine; Health Psychology; Psychosocial Intervention; People Who Inject Drugs
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Volitional help sheet
  Interventions: Behavioral: Volitional Help Sheet
- Control (No Intervention): Short Zimbardo's time perspective inventory (Orosz et al. 2017)

INTERVENTIONS:
Behavioral: Volitional Help Sheet — This brief intervention will last around 20 minutes. The participants and the researcher will read through the list of real-life solutions the participants might find applicable to them. They will then read through the list of situations one by one. The participant will draw a coloured line between the situation and the solution which seems more appropriate to them. The volitional help sheet helps create implementation intentions, which are self-regulatory strategies taking the form of "if-then" plans (i.e. situation-solution plan).
  Arms: Intervention

SUMMARY:
The study evaluates the use of implementation intentions to increase self-efficacy and reduce injecting risk behaviour in a sample of injecting drug users on treatment for hepatitis C (HCV). The overall aim is to reduce HCV reinfection rates. The primary objective is to identify lower injecting risk behaviour scores in patients on treatment for hepatitis C receiving the psychosocial intervention compared to the same patient group assigned to the control group.

DETAILED DESCRIPTION:
The intervention will entail completing a volitional help sheet.This will create implementation intentions, which are self-regulatory strategies taking the form of "if-then" plans (i.e. situation-solution plan).

Injecting risk behaviour scores and self-efficacy scores will be analysed for differences between intervention and control groups.

To control for contact-time with the researchers, participants in the control group will spend approximately 20 minutes with the researcher exploring Zimbardo's time perspective constructs (ZTPI, Zimbardo & Boyd, 1999) and completing the short Zimbardo's time perspective inventory (Orosz et al. 2017). The inventory was selected because the cognitive processes involved in accessing time constructs will also be activated in the intervention group for the planning of coping strategies and goal achievement during future injecting risk situations.

The study also aims:

* To assess the variability in injecting risk behaviour as explained by subjective norms, social connectedness and group identification constructs;
* To assess the variability in intervention effectiveness as explained by changes in mental health, illness perception subjective norms, social connectedness, and group identification.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female. (Over 18 years of age);
* Chronic HCV positive infection;
* Current illicit drug use established through participants' self-report;
* Current HCV treatment provided by the NHS;
* Informed consent, agreeing to study and monitoring criteria;
* English-speaking.

Exclusion Criteria:

* Inability to provide informed consent;
* Aggressive or violent behaviour;
* Not currently receiving HCV treatment;
* Inability to communicate in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
Injecting Risk Behaviour | 4 weeks
  Self-reported injecting risk behaviour over the past 4 weeks. Seventeen items scored 1-4 (1 frequently, 4 never)
Self-Efficacy | 4 weeks
  Self-reported confidence in one's own ability to refuse sharing of injecting equipment and use of old injecting equipment. Fifteen items scored 1-7 (1 high confidence, 7 low confidence)

SECONDARY OUTCOMES:
Subjective Norms | Up to 4 weeks
  Self-reported social norms of individual's injecting network. Four items scored 1-7 (1 strong acceptance of sharing equipment, 7 no acceptance of sharing equipment).
Social Connectedness | Up to 8 weeks
  Self-reported perceived social connectedness to general society. Eight items scored 1-6 (1 low connectedness, 6 high connectedness)
Group Identification | Up to 8 weeks
  Self-reported perceived identification with family group and injecting group. Eight items scored 1-7 (1 high identification, 7 low identification).
Depression | 2 weeks
  Self-reported depressive symptoms over the past 2 weeks. Nine items scored 0-3 (0 no symptoms, 3 depressive symptoms)
Anxiety | 2 weeks
  Self-reported depressive symptoms over the past 2 weeks. Nine items scored 0-3 (0 no symptoms, 3 depressive symptoms)
Post traumatic stress disorder | 1 month
  Self-reported trauma-induced stress symptoms over the past month. Five items scored Yes/No.
Working alliance | Treatment duration (12 weeks)
  Self-reported therapeutic alliance with provider of hepatitis C treatment care over treatment duration. Eight items scored 1-5 (1 poor alliance, 5 excellent alliance).
Illness perception | Up to 8 weeks
  Self-reported perception of hepatitis C as an illness. Eight items scored 1-10 (1 no impact on quality of life, 10 high impact on quality of life).

CONTACTS AND LOCATIONS:
Locations (1):
- Cairn Centre Needle Exchange, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: No